CLINICAL TRIAL: NCT01647386
Title: Pilot Study Using Radiostereometric Analysis (RSA) to Evaluate the Fixation of the Tibial Components in the DePuy M.B.T. Revision Knee System
Status: Completed | Type: Observational
Sponsor: Michael Dunbar (Other)
Responsible Party: Sponsor-Investigator, Michael Dunbar, Orthopedic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: DEP_MBT
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Revision Total Knee Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MBT Revision Component

SUMMARY:
Motivated by the growing number of revision total knee arthroplasty (TKAs) and the interest among surgeons to quantify the effectiveness of specific implant designs, the goal of the current project is to use Radiostereometric Analysis (RSA) to provide conclusive and clinically relevant results on fixation of the tibial component with the DePuy M.B.T. Revision TKA system using Metaphyseal Sleeves.

Does the tibial component of the M.B.T. Revision Knee System achieve adequate fixation to the underlying bone (proximal tibia) as measured by migration? • Null Hypothesis: The maximum total point motion (MTPM) value of migration of the M.B.T. Revision Knee System component between postoperative years one and two does not exceed 0.2 mm indicating adequate long-term fixation at the bone-implant interface.

• Alternative Hypothesis: The MTPM value of migration of the M.B.T. Revision Knee System component between postoperative years one and two does exceed 0.2 mm indicating inadequate long-term fixation at the bone-implant interface.

b) In what proportion of patients is adequate fixation achieved?

ELIGIBILITY:
Inclusion Criteria:

* Revision TKA is indicated and it is the opinion of the investigator that the PFC Sigma M.B.T. Tibial component with metaphyseal sleeves and a stem is a suitable treatment
* Contained bone defects in the proximal tibia that allow for contiguous contact between metaphyseal sleeves and cortical bone
* Use of tibial stem
* Ability to give informed consent

Exclusion Criteria:

* Revision TKA due to infection
* Patellar revision only
* Polyethylene liner exchange only
* Revision requiring hinged TKA
* Uncontained defects in the proximal tibia that preclude contiguous contact between metaphyseal sleeves and cortical bone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Failed primary TKR
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Implant Migration | 2 years

SECONDARY OUTCOMES:
BMD | 2 years

OTHER OUTCOMES:
Health outcome questionnaire | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunbar, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada